CLINICAL TRIAL: NCT02089529
Title: Treatment of Axial Spondyloarthritis With Reduced Doses of NSAIDs: Application of Pharmacotherapeutic Conditioning in Clinical Practice.
Brief Title: Treatment of Axial Spondyloarthritis With Reduced Doses of NSAIDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2010/2528(REK); 2013-000098-65 (EudraCT Number)
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial Spondyloarthritis; Pain; NSAIDs; Placebo; Placebo intervention; Stress; Conditioning
MeSH Terms: conditions — Axial Spondyloarthritis; Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Ibuprofen/Ibumetin (Active Comparator): Ibumetin is administrated. Intervention: No information about the effect.
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Placebo is administrated. Intervention: No information about the effect.
  Interventions: Drug: Placebo
- Ibuprofen/Ibumetin+positive information (Active Comparator): Ibumetin is administrated. Intervention: The patient receive written information that the capsule is Ibumetin.
  Interventions: Drug: Ibuprofen
- Placebo+positive information (Placebo Comparator): Placebo is administrated. Intervention:The patient receive written information that the capsule is Ibumetin.
  Interventions: Drug: Placebo
- Ibuprofen/Ibumetin+neutral information (Active Comparator): Ibumetin is administrated. Intervention: The patient receive written information that the capsule is Ibumetin.
  Interventions: Drug: Ibuprofen
- Placebo+neutral information (Placebo Comparator): Placebo is administrated. Intervention:The patients receive information that the capsule is placebo.
  Interventions: Drug: Placebo
- Control (No Intervention): Control condition

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen/Ibumetin with no information, positive information and neutral information
  Other Names: Ibumetin
  Arms: Ibuprofen/Ibumetin; Ibuprofen/Ibumetin+neutral information; Ibuprofen/Ibumetin+positive information
Drug: Placebo — Placebo with no information, positive information and neutral information
  Arms: Placebo; Placebo+neutral information; Placebo+positive information

SUMMARY:
The following study investigates the role of information/expectancies in the response to Ibumetin and placebo.

The study is a double-blind randomized controlled trial with crossover, within subjects repeated measurements. The symptoms are measured by questionnaires. 40 patients will be included in the study. The administrated drug is Ibumetin 400 mg.

The study does not require patients to meet in the clinic. Patients will be instructed in how to report pain, tension and nervousness via mobile phone (Checkware AS, Trondheim, Norway).Three days a week for 12 weeks the patients are instructed to report at 0900 AM, and thereafter at 0910, 1100, 1300, 1500, 1700, and 1900 hrs each study day. At these times the patients will receive a sms where they are instructed to immediately rate their pain and stress level and report back.

DETAILED DESCRIPTION:
The study is a double-blind randomized controlled trial with crossover, within subjects repeated measurements. The symptoms are measured by questionnaires. 40 patients will be included in the study. Patients are recruited via the Department of Rheumatology, UNN. The patient group is selected because they respond well to NSAIDs. Since the patients can participate while being at home it is not a requirement to live in Tromsø.

When the patients are recruited their normal treatment plan is examined. This includes both their prescript treatment from the patient's physicians and also non-prescript substances, such as herbal medicine. If these drugs or substances inflict with the study treatment plan, the patients will be excluded. The patient will follow the study treatment plan on study days only, which is three days during the week. During the study days the patients will be required to abstain from any other substances that can influence the treatment, such as alcohol, both prescription and nonprescription drugs and herbal medicine. After 19:00 the study day is over and other medication can be taken. On the non-study days the patients can follow their normal treatment plan, but if the following day is a study day, no medication can be consumed after 21:00.

The patients can at any time withdraw from the study. A patient who withdraws from the study will not be replaced.

Data collection

The study does not require patients to meet in the clinic. The patients can be at home, at work or performing their daily routines as they participate. Information about the procedures of self-administration will either be given to the patients in written form through mail or in person by the experimenter. Patients will be instructed in how to report pain, tension and nervousness via mobile phone (Checkware AS, Trondheim, Norway). Data from the sms is automatically saved in a database administrated by Checkware AS and the research team. The patient's phone number is connected to a patient ID number in the database. The patients name is connected to the same identification number in a different document safely secured on a different hard disk.

Submission via sms has the advantage that most people have their mobile phone with them at most times. Additionally, the time of recording is registered, which cannot be reliably done via paper and pencil recordings. Three days a week for 12 weeks the patients are instructed to report at 0900 AM, and thereafter at 0910, 1100, 1300, 1500, 1700, and 1900 hrs each study day. At these times the patients will receive a sms where they are instructed to immediately rate their pain and stress level and report back. If they do not report within 10 minutes they will receive a new sms as a reminder. Patients will also be instructed to send in the SF-36 and the Fear of Pain Questionnaire at the inclusion of the study, midway and at the final day.

Endpoints:

Primary endpoints: pain intensity and pain unpleasantness are measured by numerical rating scales (NRS) via sms. Perceived health related quality of life measured with Sort Form (36) Health Survey in Norwegian translation [22]. Secondary endpoints: tension and nervousness measured on NRS via sms. Fear of pain measured by The Fear of Pain Questionnaire III in Norwegian translation [23].

Questionnaires Short Form (36) Health Survey The Short Form (36) Health Survey (SF(36)) is a standardized and validated self-report questionnaire that assesses how patient perceive their own health. It is normally used to measure health status in clinical studies. The present study will use a Norwegian translation of the questionnaire.

The Fear of Pain Questionnaire III The Fear of Pain Questionnaire III (FPQ-III) is a standardized and validated self-report questionnaire that assesses fear of pain. It contains of 30 items involving three subscales: Severe pain, minor pain and medical pain. Each item is rated on a five-point Likert scale, were 1=no fear and 5=extreme fear. The present study will use a Norwegian translation of the FPQ-III.

Pharmaceutical control and placebo Kragerø Tablettproduksjon (in Kragerø, Norway) will be responsible for the pharmaceutical control. The administrated drug is Ibumetin 400 mg (http://www.felleskatalogen.no/medisin/ibumetin-takeda-nycomed-559938). The placebo is capsules containing sugar spheres produced by Kragerø Tablettproduksjon. To secure that the Ibumetin and the placebo looks identical; the Ibumetin will be purchased by Kragerø Tablettproduksjon from the producer of Ibumetin, Takeda Nycomed, and then sealed in identical capsules as the placebo.

Kragerø Tablettproduksjon will label and pack the entire 12 week treatment. The treatment dose for each day will be put in separate containers. The containers will be marked with a number from 1-35 representing the specific treatment day.

The treatment order is different for each patient, and Kragerø Tablettproduksjon has received the treatment order for every patient from the Department of Psychology, UiT.

Randomization and blinding:

When the patients have been enrolled they receive an ID-number. To secure double blinding an independent researcher at the Department of Psychology, who is not involved in the study, will administer the ID-number distribution using www.random.org. The ID-number is also linked to a specific order of treatment and the order of treatment is different for every patient. The lists (1) linking each patient to their ID-number and (2) linking the treatment order to the different ID-numbers will be filed separately from other study information and not be released to the conductors. However, if circumstance requires, such as severe side effects resulting in hospital admission or death (see below), the blinding for the specific patient or patients will be released to the conductors.

Design:

A 2 drug (Ibumetin and placebo) x 3 information (no information, positive, neutral) within subjects repeated measures (pre-test, 6 post-tests) design will be conducted. All patients will be tested in all conditions.

Condition 1: Baseline: Pain and stress registered, Ibumetin placebo not administrated.

Condition 2: Ibumetin: Ibumetin administrated. No information about the effect. Condition 3: Placebo: Placebo administrated. No information about the effect.

Condition 4: Ibumetin + Positive Information: Ibumetin administrated. The patients receive written information that the capsule is Ibumetin.

Condition 5: Placebo + Positive Information: Placebo administrated. The patients receive written information that the capsule is Ibumetin.

Condition 6: Ibumetin + Neutral Information: Ibumetin administrated. The patients receive written information that the capsule is placebo.

Condition 7: Placebo + Neutral Information: Placebo administrated. The patients receive written information that the capsule is placebo.

Procedure:

Patients that have been enrolled and have signed the informed consent are informed about the purpose of the experiment and the procedures. Patients will orally self-administer 4 capsules containing Ibumetin 400 mg or identical looking capsules with placebo every Monday, Wednesday and Friday morning for 12 consecutive weeks in their home environment. The administrated treatment dose of Ibumetin is normal in treatment of pain in patients with Axial SpA. The patients will report their score on the outcome variables via mobile phone in accordance with the schedule mentioned above. The seven conditions are presented five times to each participant, for 35 days, with one workday between each condition. For the first seven study days, each condition is run once, for study days eight to 14 each condition is run once, etc. Thus, the 35 study days are comprised of five blocks of seven study days, in which all conditions are presented. The order of presentations of the conditions is random within each block and is different in all participants. The subjects are allowed to take non-study medicine on non-study days and after 1900 hours on study days, but not after 2100 hours if the following day is a study day. The SF-36 and FOP questionnaires are filled in upon inclusion in the study, and again after study days 17 and 35.

The participants will receive the capsules in Nolato 50 ml/34 mm containers (box: Art.no C112863 Cerbo Classic 50 ml white, lid: Art.nr.: C112820 Cerbo Classic SC 34 white) with all relevant information . The patients will also be encouraged to contact the conductors by phone if they have any questions or worries.

The patients will be informed that it is necessary to follow the treatment protocol precisely as described, and that any variance will compromise the study. The patients will be equipped with a "study journal". In the study journal the patients have to register what time they take their treatment and if they consume all the capsules. The patients also have to register what substances they consume on non-study days. The study journal will also have a note section. In this section the patients can note what they think of the treatment, how they feel, if they experience any side effects, if they experience any new medical incidences or if they feel stressed and uncomfortable. They also have to register if they have followed the treatment plan as requested and if they have answered the questionnaires. When the study is completed the patients will be asked if they did follow the treatment protocol exactly, and encouraged to be truthful. If they report any mistakes or variance, it will be noted and included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with radiographic Axial Spondyloarthritis, also called Ankylosing Spondylitis, OR
* Patients must have been diagnosed with non-radiographic Axial Spondyloarthritis with a positive magnetic resonance (MR).
* Patients must have been successfully treated with NSAIDs for at least three months
* Patients must be above 20 years old
* Patients must satisfy the Norwegian Summary of Product Characteristics (SPC) for Ibumetin 400 mg
* All patients must sign a consent form describing that they will receive placebo during the study period. The Informed Consent Form and The Data Release Form must be signed before inclusion in the studies.

Exclusion Criteria:

* Patients cannot participate in other clinical studies parallel to the current study. Previous study participations must be completed more than one year, prior to participating in the current study.
* Patients not satisfying the Norwegian Summary of Product Characteristics (SPC) for Ibumetin 400 mg:
* Patients who previously have experienced allergic reactions to NSAIDs
* Patients with previous or currant ulcers and/or gastrointestinal conditions - or bleeding
* Patients with previous or currant cardiovascular conditions, or have experienced cardiovascular episodes
* Patients with previous or currant renal failure
* Patients with acetaminophen - or NSAID-induced asthma, urticarial or rhinitic
* Patients with previous or current other serious conditions apart from rheumatoid arthritis
* Female patients trying to or having trouble getting pregnant cannot participate in the study
* Pregnant and/or nursing patients cannot participate in the study
* Patients on a treatment plan with Prednisolon
* Patients on a treatment plan with substances inflicting with Ibumetin. All substances will be investigated on www.interaksjoner.no

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in level of pain | up to 12 weeks

SECONDARY OUTCOMES:
Change in level of stress and nervousness | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gunnstein Bakland, MD, phd, Principal Investigator — UNN; Magne Arve Flaten, psycol, phd, Study Director — UIT
Locations (1):
- University Hospital of Northen Norway, Tromsø, Tromsø, Norway